CLINICAL TRIAL: NCT03870100
Title: Use the Protocol Title. The Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study Following A Single Subcutaneous Injection of SHR-1222 in Healthy Subjects
Brief Title: The PK/PD Study of A Single Subcutaneous Injection of SHR-1222 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1222-101
Record Dates: First submitted 2019-02-25; First posted 2019-03-11 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): A single subcutaneous injection of SHR-1222 dose 1 versus placebo
  Interventions: Drug: SHR-1222; Drug: Placebo
- Cohort 2 (Experimental): A single subcutaneous injection of SHR-1222 dose 2 versus placebo
  Interventions: Drug: SHR-1222; Drug: Placebo
- Cohort 3 (Experimental): A single subcutaneous injection of SHR-1222 dose 3 versus placebo
  Interventions: Drug: SHR-1222; Drug: Placebo
- Cohort 4 (Experimental): A single subcutaneous injection of SHR-1222 dose 4 versus placebo
  Interventions: Drug: SHR-1222; Drug: Placebo
- Cohort 5 (Experimental): A single subcutaneous injection of SHR-1222 dose 5 versus placebo
  Interventions: Drug: SHR-1222; Drug: Placebo

INTERVENTIONS:
Drug: SHR-1222 — Pharmaceutical form: water injection Route of administration: subcutaneous
Drug: Placebo — Pharmaceutical form: water injection Route of administration: subcutaneous

SUMMARY:
This is a Single Center, Randomized, Double-Blind, Dose Escalation, Placebo Parallel Controlled PhaseⅠClinical study to Evaluate the Safety, Tolerability and Pharmacokinetics, Pharmacodynamics with A Single Subcutaneous Injection of SHR-1222 in Healthy Subjects.

The primary objective of this study is to investigate the safety and tolerability of a range of subcutaneous SHR-1222 in healthy subjects. Secondary objectives are to determine the pharmacokinetics (PK) and pharmacodynamics(PD) profile of SHR-1222 in healthy subjects including assessment of immunogenicity.

DETAILED DESCRIPTION:
50 adult healthy subjects with 5 dose groups will be enrolled in the study, including six subjects in the lowest dose group, four of whom received the SHR-1209 and two of whom received the placebo. The other three groups have 11 subjects in each group, 9 administered SHR-1222 and 2 administered placebo. The primary endpoint is the Safety and Tolerability : adverse events, vital signs, physical examination, laboratory examination, 12 lead electrocardiogram, injection site reactions, etc.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Male or postmenopausal female;
* Age ≥45 and ≤59 years old;
* The body mass index (BMI) ≥18.5kg/m2 and ≤28 kg/m2;
* T value of areal bone mineral density on any lumbar spine (L1-L4) or collum femoris>-2.5 and <-1;
* The comprehensive physical examination is eligible or slightly abnormal but the researchers determine no clinical implication;
* No smoking, alcohol or drugs abuse.

Exclusion Criteria:

* Any disease affecting bone metabolism;
* Past medical history of cerebral infarction or cerebral arterial thrombosis;
* Past medical history of myocardial infarction;
* Administration of the following drugs within 6m: Hormone replacement therapy, Calcitonin Parathyroid hormone (or any derivative), Supplemental Vitamin D>1,000 IU/day, Glucocorticosteroids (inhaled or topical corticosteroids administered more than 2 weeks before the enrollment date are allowed), Anabolic steroids, Calcitriol and available analogues, thiazide diuretics;
* Administration of the following drugs within 12m: Bisphosphonates, Fluoride for osteoporosis;
* A bone fracture within the previous 6 months;
* A lumbar spine L1-L4 or femoral neck T-score ≤-2.5;
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or gamma pancreatic acyl transferase (GGT) or total bilirubin, more than 1.5 x ULN during screening;
* 3 months prior to screening involved in any drug clinical subjects;
* Subjects determined by the researchers have any food, dietary supplement or drugs that affect SHR-1222 absorption, distribution, metabolism and excretion in 4 weeks prior to screening or within 5 half-lives;
* Serious infection, trauma or major surgery in 4 weeks prior to screening;
* A surgery plan during the study;
* Blood donation and transfusion in 3 months prior to screening;
* Unstable thyroid dysfunction in 6 months prior to screening;
* Human immunodeficiency virus antibody (HIV-ab), syphilis serological examination, hepatitis b virus surface antigen (HBsAg), hepatitis c virus antibody (HCV-ab) were positive;
* Intolerant to venous blood collection;
* A clinical history of drug allergy or a history of atopic allergic diseases (asthma, urticaria, eczema dermatitis) or a known allergy to experimental or similar
* Subjects with any other situation should not be involved, which determined by the researchers.

Ages: 45 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Number & proportion of subjects with adverse events [Time Frame: dose administration to 85 days after dose administration] Safety and Tolerance: Number & proportion of subjects with adverse events | Dose administration to 85 days after dose administration

SECONDARY OUTCOMES:
Assessment of PK parameter-time to maximum concentration (Tmax) | Pre-dose to 85 days after dose administration
Assessment of PK parameter-maximum concentration (Cmax) | Pre-dose to 85 days after dose administration
Assessment of PK parameter-area under curve (AUC) | Pre-dose to 85 days after dose administration
Assessment of PD parameter-change in serum C-telopeptide (sCTx) from baseline | Pre-dose to 85 days after dose administration
Assessment of PD parameter-change in aminoterminal propeptide type-1 procollagen (P1NP) from baseline | Pre-dose to 85 days after dose administration
Assessment of PD parameter-change in osteocalcin from baseline | Pre-dose to 85 days after dose administration
Assessment of PD parameter-change in bone-specific alkaline phosphatase (BSAP) from baseline | Pre-dose to 85 days after dose administration
Assessment of PD parameter-change in areal bone mineral density of lumbar spine (L1-L4 mean T value) from baseline | Pre-dose to 85 days after dose administration
  by dualenergy X-ray absorptiometry
Assessment of PD parameter-change in areal bone mineral density of collum femoris (T value) from baseline | Pre-dose to 85 days after dose administration
  by dualenergy X-ray absorptiometry
Assessment of PD parameter-change in volumetric bone mineral density of lumbar spine (L1-L4 mean T value) from baseline | Pre-dose to 85 days after dose administration
  by quantitative computed tomography
Assessment of PD parameter-change in volumetric bone mineral density of collum femoris (T value) from baseline | Pre-dose to 85 days after dose administration
  by quantitative computed tomography
Antidrug antibody concentration | Pre-dose to 85 days after dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguang Zhou, MD, Principal Investigator — 2nd Xiangya Hospital of Central South University
Locations (1):
- 2nd Xiangya Hospital of Central South University, Changsha, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dai Z, Fang P, Yan X, Zhu R, Feng Q, Yan Q, Yang L, Fan X, Xie Y, Zhuang L, Feng S, Liu Y, Zhong S, Yang Z, Sheng Z, Zhou Z. Single Dose of SHR-1222, a Sclerostin Monoclonal Antibody, in Healthy Men and Postmenopausal Women With Low Bone Mass: A Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation, Phase I Study. Front Pharmacol. 2021 Oct 20;12:770073. doi: 10.3389/fphar.2021.770073. eCollection 2021. PMID 34744750